CLINICAL TRIAL: NCT04353596
Title: Stopping ACE-inhibitors in COVID-19: A Randomized Controlled Trial
Brief Title: Stopping ACE-inhibitors in COVID-19
Acronym: ACEI-COVID
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Collaborators: Ludwig-Maximilians - University of Munich (Other); Deutsches Zentrum für Herz-Kreislauf-Forschung (DZHK) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EudraCT 2020-001206-35
Record Dates: First submitted 2020-04-14; First posted 2020-04-20 (Actual); Results first posted 2022-09-13 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2021-02

CONDITIONS: SARS-CoV-2; COVID-19
Keywords: ACE-inhibitors; RAS system; angiotensin receptor blockers; SARS-CoV-2; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Angiotensin-Converting Enzyme Inhibitors; Angiotensin Receptor Antagonists

STUDY DESIGN:
Intervention Model Description: open-label, randomized design
Who Masked: Outcomes Assessor
Masking Description: unmasked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Stopping/replacing ACEI/ARB (Experimental): Chronic treatment with ACEI or ARB will be stopped or replaced.
  Interventions: Drug: ACE inhibitor, angiotensin receptor blocker
- Control (No Intervention): No intervention, which means further treatment with ACEI or ARB.

INTERVENTIONS:
Drug: ACE inhibitor, angiotensin receptor blocker — In patients randomized to stopping / replacing ACEI or ARB, it may be necessary to switch to another drug without direct effect on the RAS system. In patients, randomized to continuation, it may be needed to stop ACEI or ARB (e.g. hypotension with beginning sepsis) irrespective of the study.
  Arms: Stopping/replacing ACEI/ARB

SUMMARY:
ACEI-COVID-19 is a multicenter, randomized trial testing the hypothesis that stopping/replacing chronic treatment with ACE-inhibitors (ACEI) or angiotensin receptor blockers (ARB) improves outcomes in symptomatic SARS-CoV2-infected patients

DETAILED DESCRIPTION:
The COVID-19 pandemic currently poses unprecedented challenges to the health systems of all countries. Experimental studies show that the SARS-CoV2 virus enters human cells via the angiotensin converting enzyme II receptor 2 (ACE2). ACE inhibitors (ACEI) and angiotensin receptor blockers (ARB) can lead to an increase in the expression of ACE2. Therefore, there is concern that in patients treated with ACEI or ARB, the absorption of the virus is facilitated, thereby accelerating its spread in the body.

ACEI-COVID tests the hypothesis that stopping chronic ACEI / ARB therapy in SARS-CoV2-infected patients improves outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients competent to make a decision
* Proven and symptomatic SARS-CoV2 infection ≤ 5 days
* Patient age ≥ 18 years
* Provided written informed consent
* Chronic (≥ 1 month) ACEI/ARB therapy for treatment of arterial hypertension, diabetes mellitus, heart failure or coronary artery disease
* Stable hemodynamic conditions allowing to stop or continue treatment with ACEI/ARB (systolic blood pressure ≤180mmHg)

Exclusion Criteria:

* Women capable of bearing children as well as pregnant and breastfeeding women
* Participant in another interventional trail
* At screening visit, no oral medication intake possible
* Advanced heart failure NYHA Stage III-IV
* Left ventricular ejection fraction <30% or NTproBNP ≥600pg/mL in case of clinical signs of heart failure
* Acute coronary syndrome ≤ 3 months
* Severe arterial hypertension (concomitant use of more than 4 different antihypertensive drug classes)
* Acute respiratory distress syndrome with need for mechanical ventilation
* Patients who at not capable of home blood pressure monitoring
* Patients who cannot be switched to an alternative medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2021-02-16 (Actual); Study Completion 2021-02-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (31):
- Austria (14):
  - Medical University Innsbruck, University Hospital of Internal Medicine III, Innsbruck, Tyrol
  - Medical University of Graz, Graz
  - Landeskrankenhaus Hall, Hall in Tirol
  - Medical University Innsbruck, Intensive Care and Emergency Medicine Department, Innsbruck
  - Medical University Innsbruck, University Hospital of Internal Medicine II, Innsbruck
  - Medical University Innsbruck, University Hospital of Internal Medicine IV, Innsbruck
  - Medical University Innsbruck, University Hospital of Internal Medicine I, Innsbruck
  - Medical University Innsbruck, University Hospital of Internal Medicine V, Innsbruck
  - Klinikum Klagenfurt, Klagenfurt
  - Bezirkskrankenhaus Kufstein, Kufstein
  - Klinikum Lienz, Lienz
  - Bezirkskrankenhaus St. Johann, Sankt Johann in Tirol
  - Bezirkskrankenhaus Schwaz, Schwaz
  - Krankenhaus St. Vinzenz Zams, Zams
- Germany (17):
  - LMU Klinikum, Medizinische Klinik I, Munich, Bavaria
  - University Hospital Aachen, Aachen
  - University Hospital Augsburg, Augsburg
  - Asklepios Stadtklinik Bad Tölz, Bad Tölz
  - Klinikum Dachau, Dachau
  - University Hospital Erlangen, Erlangen
  - University Hospital Essen, Essen
  - University of Freiburg, Freiburg im Breisgau
  - Klinikum Memmingen, Memmingen
  - LMU Klinikum, Medizinische Klinik III, Munich
  - LMU Klinikum, Medizinische Klinik II, Munich
  - LMU Klinikum, Medizinische Klinik IV, Munich
  - München Klinik Bogenhausen und Schwabing, Munich
  - Rotkreuzklinikum Munich, Munich
  - Krankenhaus Mühldorf, Mühldorf
  - Klinikum Rosenheim, Rosenheim
  - Krankenhaus Weiden, Weiden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bauer A, Schreinlechner M, Sappler N, Dolejsi T, Tilg H, Aulinger BA, Weiss G, Bellmann-Weiler R, Adolf C, Wolf D, Pirklbauer M, Graziadei I, Ganzer H, von Bary C, May AE, Woll E, von Scheidt W, Rassaf T, Duerschmied D, Brenner C, Kaab S, Metzler B, Joannidis M, Kain HU, Kaiser N, Schwinger R, Witzenbichler B, Alber H, Straube F, Hartmann N, Achenbach S, von Bergwelt-Baildon M, von Stulpnagel L, Schoenherr S, Forer L, Embacher-Aichhorn S, Mansmann U, Rizas KD, Massberg S; ACEI-COVID investigators. Discontinuation versus continuation of renin-angiotensin-system inhibitors in COVID-19 (ACEI-COVID): a prospective, parallel group, randomised, controlled, open-label trial. Lancet Respir Med. 2021 Aug;9(8):863-872. doi: 10.1016/S2213-2600(21)00214-9. Epub 2021 Jun 11. PMID 34126053

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between April 20, 2020, and Jan 20, 2021, 204 participants were randomly assigned to discontinuation (n=109) or continuation (n=107) of RAS inhibition, at 35 centres, including 19 university clinics and 16 large referral hospitals, in Austria and Germany.
Pre-assignment Details: Of 2301 patients, who were assessed for eligibility, 216 underwent randomization. 1921 were excluded due violation of inclusion or exclusion criteria.
Groups:
- Discontinuation Group: Discontinuation of chronic ACEI or ARB pretreatment
- Continuation Group: Continuation of chronic ACEI or ARB pretreatment
Period: Overall Study
Arm/Group | Discontinuation Group | Continuation Group
Started | 109 | 107
Per Protocol | 104 | 100
Completed | 104 | 100
Not Completed | 5 | 7
Not completed — Protocol Violation | 4 | 4
Not completed — no evidence of recent SARS-CoV-2 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Discontinuation Group: Chronic pretreatment with ACEI or ARB will be stopped or replaced.
  Substitution with an alternative substance class was at the discretion of the treating physician
- Continuation Group: No intervention, which means further treatment with ACEI or ARB. In patients, randomized to continuation, it may be needed to stop ACEI or ARB (e.g. hypotension with beginning sepsis) irrespective of the study.
- Total: Total of all reporting groups
Arm/Group | Discontinuation Group | Continuation Group | Total
Number analyzed (Participants) | 104 | 100 | 204
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 74 [62 to 80] | 75 [69 to 80] | 75 [66 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 36 | 75
  Male | 65 | 64 | 129
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 104 | 100 | 204
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Austria | 59 | 57 | 116
  Germany | 45 | 43 | 88
BMI [Median (Inter-Quartile Range); unit: "kg per m^2"] | 28 [25.4 to 31.3] | 27.4 [25.4 to 29.4] | 27.6 [25.5 to 30.5]
Hypertension [Count of Participants; unit: Participants] | 100 | 99 | 199
Current Smoker [Count of Participants; unit: Participants] | 6 | 99 | 105
Dyslipidaemia [Count of Participants; unit: Participants] | 38 | 48 | 86
Diabetes [Count of Participants; unit: Participants] | 30 | 37 | 67
Coronary artery disease [Count of Participants; unit: Participants] | 22 | 23 | 45
Heart failure [Count of Participants; unit: Participants] | 12 | 6 | 18
Chronic obstructive pulmonary disease [Count of Participants; unit: Participants] | 10 | 22 | 32
Atrial fibrillation [Count of Participants; unit: Participants] | 18 | 17 | 35
Malignant disease [Count of Participants; unit: Participants] | 7 | 13 | 20
Kidney disease [Count of Participants; unit: Participants] | 16 | 21 | 37
History of stroke [Count of Participants; unit: Participants] | 8 | 5 | 13
Angiotensin-converting enzyme inhibitor [Count of Participants; unit: Participants] | 57 | 58 | 115
Angiotensin II receptor blocker [Count of Participants; unit: Participants] | 47 | 42 | 89

OUTCOME MEASURES:

1. Primary Outcome: Composite of the Maximum Sequential Organ Failure Assessment (SOFA) Score and Death Within 30 Days
Description: The score is calculated from six different components, each of which reflects the status of an organ system, including respiratory function, cardiovascular integrity, liver function, coagulation, renal function and neurological status. The score can range from 0 (best) to 24 (worst). In case of death, the patient was by definition assigned the maximum value of 24. Outpatients were assigned a value of 0 or 24 (in the case of death).
Time Frame: 30 days
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Discontinuation Group: Discontinuation of ACEI or ARB therapy
- Continuation Group: Continuation of ACEI or ARB therapy
Arm/Group | Discontinuation Group | Continuation Group
Number analyzed (Participants) | 104 | 100
score on a scale | 0 [0 to 2] | 1 [0 to 3]

2. Primary Outcome: Composite of Admission to an Intensive Care Unit (ICU), the Use of Mechanical Ventilation, or All-cause Death
Description: Composite of admission to ICU, mechanical ventilation, and death
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Discontinuation Group | Continuation Group
Number analyzed (Participants) | 104 | 100
Participants | 21 | 26

3. Secondary Outcome: Mean of Sequential Organ Failure Assessment (SOFA) Score
Description: minimum score is 0, maximum score is 24; higher score indicates poor outcome (death-adjusted)
Time Frame: 30 days
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Discontinuation Group | Continuation Group
Number analyzed (Participants) | 104 | 100
score on a scale | 0 [0 to 0.31] | 0.12 [0 to 0.78]

4. Secondary Outcome: Rates of Non-invasive Ventilation
Description: Number of Participants with Non-invasive Ventilation
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Discontinuation Group | Continuation Group
Number analyzed (Participants) | 104 | 100
Participants | 19 | 14

5. Secondary Outcome: Rates of Renal Replacement Therapies
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Discontinuation Group | Continuation Group
Number analyzed (Participants) | 104 | 100
Participants | 0 | 1

6. Secondary Outcome: Number of Patients With Systolic/Diastolic Blood Pressure > 180/120 mmHg
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Discontinuation Group | Continuation Group
Number analyzed (Participants) | 104 | 100
Participants | 7 | 7

7. Secondary Outcome: Hospitalisation Due to Cardiac Decompensation
Description: with causal relationship to stopping of ACEI/ARB therapy
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Discontinuation Group | Continuation Group
Number analyzed (Participants) | 104 | 100
Participants | 0 | 0

8. Secondary Outcome: Rates of Mechanical Ventilation
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Discontinuation Group | Continuation Group
Number analyzed (Participants) | 104 | 100
Participants | 10 | 8

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Discontinuation Group | Continuation Group
All-Cause Mortality (participants affected / at risk) | 8/104 | 12/100
Serious Adverse Events (participants affected / at risk) | 25/104 | 28/100
Other Adverse Events (participants affected / at risk) | 13/104 | 7/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Discontinuation Group (N=104) | Continuation Group (N=100)
Worsening of respiratory function (Respiratory, thoracic and mediastinal disorders) | 21 | 24
Ischemic events (Cardiac disorders) | 0 | 2
Urinary tract infection (Renal and urinary disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Worsening of general condition (Infections and infestations) | 2 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Discontinuation Group (N=104) | Continuation Group (N=100)
Worsening of respiratory function (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Urinary tract infection (Renal and urinary disorders) | 2 | 0
Elevation of creatinine (Renal and urinary disorders) | 0 | 1
Hypertension (Vascular disorders) | 2 | 2
Worsening of general condition (Infections and infestations) | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-06): https://cdn.clinicaltrials.gov/large-docs/96/NCT04353596/Prot_SAP_000.pdf